CLINICAL TRIAL: NCT05415072
Title: A Phase I/II, Multi-center, Open Label Study of DYP688 in Patients With Metastatic Uveal Melanoma (MUM) and Other GNAQ/11 Mutant Melanomas
Brief Title: A Phase I/II Study of DYP688 in Patients With Metastatic Uveal Melanoma and Other GNAQ/11 Mutant Melanomas
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CDYP688A12101; 2021-003380-95 (EudraCT Number)
Record Dates: First submitted 2022-06-08; First posted 2022-06-10 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Uveal Melanoma
Keywords: Phase I/II; DYP688; melanoma; GNAQ/11 mutations; cancer; malignant melanoma; eye cancer; ocular melanoma; uveal melanoma; cutaneous melanoma; mucosal melanoma; neoplasms, eye
MeSH Terms: conditions — Uveal Melanoma; Melanoma; Neoplasms; Eye Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase I: Dose Escalation (Experimental): Patients with metastatic uveal melanoma or other GNAQ/11 mutant melanomas
  Interventions: Drug: DYP688
- Phase II: Tebe naive group (Experimental): Patients with metastatic uveal melanoma that has not received prior treatment with tebentafusp
  Interventions: Drug: DYP688
- Phase II: Tebe pre-treated (Experimental): Patients with metastatic uveal melanoma that have been previously treated with tebentafusp
  Interventions: Drug: DYP688
- Phase II: Non-uveal melanoma (Experimental): Optional Arm: To explore patients with non-uveal melanoma that harbor GNAQ or 11 mutations, based on emerging data from dose escalation
  Interventions: Drug: DYP688

INTERVENTIONS:
Drug: DYP688 — Single agent DYP688

SUMMARY:
This is a FIH, phase I/II, open label, multi-center study of DYP688 as a single agent. The purpose of this study is to characterize the safety, tolerability, and anti-tumor activity of DYP688 as a single agent in patients with metastatic uveal melanoma (MUM) and other melanomas harboring GNAQ/11 mutations.

DETAILED DESCRIPTION:
This is a First in Human (FIH), phase I/II, open label, multi-center study of DYP688 as a single agent. There will be two parts to this study: a phase I, dose escalation part followed by a phase II part. Dose escalation will be conducted in patients with MUM and other melanomas harboring GNAQ/11 mutations. Once the MTD and/or RD(s) is determined in the dose escalation part, the study may continue with a phase II part. The phase II part will be conducted in two groups of patients with MUM, a prior tebentafusp-treated group and a tebentafusp-naïve group. In addition to MUM, a third group of patients with non-uveal GNAQ/11 mutant melanomas may also be explored. This cohort may be opened based on emerging data from the dose escalation part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the dose escalation part must be ≥ 18 years of age at the time of informed consent (ICF) signature. In the phase II part, patients ≥ 12 years of age at the time of informed consent may be eligible for enrollment (not applicable in countries where enrollment is restricted by the local health authority to patients ≥ 18 years of age). Patients must have a minimum weight of 40 kg.
* ECOG performance status ≤ 1 for patients ≥ 18 years of age; Karnofsky performance status ≥ 70 for patients ≥ 16 and < 18 years of age; Lansky performance status ≥ 70 for patients ≥ 12 and < 16 years of age
* Patients must be suitable and willing to undergo study required biopsies according to the treating institution's own guidelines and requirements. If a biopsy is not medically feasible, exceptions may be considered after documented discussion with Novartis.

For all patients in Dose Escalation

* MUM: uveal melanoma with histologically or cytologically confirmed metastatic disease. Patient must be either treatment naive or have received any number of prior lines and progressed on most recent therapy
* Non-MUM: advanced cutaneous or mucosal melanoma with histologically or cytologically confirmed metastatic disease that has progressed following all standard therapies or that has no satisfactory alternative therapies and has evidence of GNAQ/11 mutation based on local data

For patients in Phase II

* Tebentafusp naïve group: Diagnosis of uveal melanoma with histologically or cytologically confirmed metastatic disease that has progressed following standard therapies or that has no satisfactory alternative therapies
* Tebentafusp pre-treated group: Diagnosis of uveal melanoma with histologically or cytologically confirmed metastatic disease. Patients must be previously treated with tebentafusp and have progressed
* Non-MUM: patients with diagnosis of cutaneous or mucosal melanomas harboring GNAQ/11 mutations based on local data, with histologically or cytologically confirmed metastatic disease that has progressed following all standard therapies or that has no satisfactory alternative therapies

Exclusion Criteria:

* Malignant disease, other than that being treated in this study.
* Active brain metastases, i.e. symptomatic brain metastases or known leptomeningeal disease.
* Evidence of active bleeding or bleeding diathesis or significant coagulopathy (including familial) or a medical condition requiring long term systemic anticoagulation that would interfere with biopsies.
* History of anaphylactic or other severe hypersensitivity / infusion reactions to ADCs or monoclonal antibodies, which in the opinion of the investigator may pose an increased risk of serious infusion reaction.
* Treatment with any of the following anti-cancer therapies prior to the first dose of study treatment within the stated timeframes:

  * 2 weeks for fluoropyrimidine therapy
  * 4 weeks for radiation therapy or limited field radiation for palliation within ≤ 2 weeks prior to the first dose of study treatment.
  * 4 weeks or ≤ 5 half-lives (whichever is shorter) for chemotherapy or biological therapy (including monoclonal antibodies) or continuous or intermittent small molecule therapeutics or any other investigational agent.
  * 6 weeks for cytotoxic agents with major delayed toxicities, such as nitrosoureas and mitomycin C.
  * 4 weeks for immuno-oncologic therapy, such as CTLA-4, PD-1, or PD-L1 antagonists.
* Clinically significant and / or uncontrolled heart disease such as congestive heart failure requiring treatment (NYHA grade ≥ 2) or clinically significant arrhythmia despite medical treatment.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Phase I (Dose Escalation): Incidence and severity of dose limiting toxicities (DLTs) during the first 28 days of treatment. | 28 days
  A DLT is defined as an adverse event or abnormal laboratory value of Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 3 assessed as unrelated to disease, disease progression, intercurrent illness, or concomitant medications that occurs within the first cycle of treatment with DYP688. Other clinically significant toxicities may be considered to be DLTs, even if not CTCAE grade 3 or higher.
Phase I (Dose Escalation): Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | 9 months
  Assessment of safety of DYP688 as a single agent
Phase I (Dose Escalation): Frequency of dose interruptions, reductions, and discontinuations | 9 months
  Assessment of tolerability of DYP688 as a single agent
Phase II: Overall Response rate (ORR) per RECIST 1.1 | 17 months
  ORR in Phase II will be evaluated by central review per RECIST 1.1.

SECONDARY OUTCOMES:
Phase I and Phase II: PK profile of DYP688 - Area under the concentration-time curve (AUC) | 26 months
  Pharmacokinetic (PK) parameters will be determined by non-compartmental methods using pharmacokinetic profile of DYP688.
Phase I and Phase II: PK profile of DYP688 - Peak concentration (Cmax) | 26 months
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of DYP688.
Phase I and Phase II: PK profile of DYP688 - Total body clearance (CL) | 26 months
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of DYP688.
Phase I and Phase II: PK profile of DYP688 - Elimination half-life | 26 months
  Pharmacokinetic parameters will be determined by non-compartmental methods using pharmacokinetic profile of DYP688.
Phase I and Phase II: Prevalence and incidence of anti-DYP688 antibodies | 26 months
  Assess of immunogenicity (IG) of DYP688 as a single agent
Phase I (Dose Escalation): Best Overall Response (BOR) per RECIST v1.1 | 9 months
  Evaluation of preliminary anti-tumor activity of DYP688 as a single agent
Phase I (Dose Escalation): Overall Response Rate (ORR) per RECIST v1.1 | 17 months
  Evaluation of preliminary anti-tumor activity of DYP688 as a single agent
Phase II: Duration of response (DoR) per RECIST v1.1 | 17 months
  Evaluation of anti-tumor activity of DYP688 as a single agent
Phase II: Progression free survival (PFS) per RECIST v1.1 | 17 months
  Evaluation of anti-tumor activity of DYP688 as a single agent
Phase II: Disease Control Rate (DCR) per RECIST v1.1 | 17 months
  Evaluation of anti-tumor activity of DYP688 as a single agent
Phase II: Overall Survival (OS) | 17 months
  Evaluation of the effect of DYP688 as a single agent on overall survival
Phase II: Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | 17 months
  Assessment of safety of DYP688 as a single agent
Phase II: Frequency of dose interruptions, reductions, and discontinuations | 17 months
  Assessment of tolerability of DYP688 as a single agent

CONTACTS AND LOCATIONS:
Locations (11):
- United States (3):
  - Massachusetts General Hospital Hematology Oncology, Boston, Massachusetts
  - Columbia University Medical Center- New York Presbyterian Onc Dept, New York, New York
  - Memorial Sloane Kettering Cancer Center MSKCC, New York, New York
- Australia (2):
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Melbourne, Victoria
- Novartis Investigative Site, Paris, France
- Germany (2):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Heidelberg
- Novartis Investigative Site, Leiden, South Holland, Netherlands
- Novartis Investigative Site, Madrid, Spain
- Novartis Investigative Site, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided